CLINICAL TRIAL: NCT05279703
Title: The Use of Epinephrine Infusion for Prophylaxis Against Maternal Hypotension During Cesarean Delivery: a Randomized Controlled Dose-finding Trial
Brief Title: Epinephrine Infusion for Prophylaxis Against Maternal Hypotension During Cesarean Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-399-2021
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Postspinal Hypotension; Cesarean Delivery; Epinephrine
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.03 mcg group (Active Comparator): epinephrine infusion will be started after subarachnoid block until 5 minutes after delivery of the baby
  Interventions: Drug: Epinephrine 0.03
- 0.02 mcg group (Active Comparator): epinephrine infusion will be started after subarachnoid block until 5 minutes after delivery of the baby
  Interventions: Drug: Epinephrin 0.02
- 0.01 mcg group (Active Comparator): epinephrine infusion will be started after subarachnoid block until 5 minutes after delivery of the baby
  Interventions: Drug: Epinephrin 0.01

INTERVENTIONS:
Drug: Epinephrine 0.03 — epinephrine infusion rate of 0.03 mcg/kg/min
  Other Names: adrenaline
  Arms: 0.03 mcg group
Drug: Epinephrin 0.02 — epinephrine infusion rate of 0.02 mcg/kg/min
  Other Names: adrenaline
  Arms: 0.02 mcg group
Drug: Epinephrin 0.01 — epinephrine infusion rate of 0.01 mcg/kg/min
  Other Names: adrenaline
  Arms: 0.01 mcg group

SUMMARY:
Maternal hypotension after spinal block is a common complication after subarachnoid block in this population. The incidence of maternal hypotension is nearly 60% when prophylactic vasopressors are not used. Therefore, it is highly recommended to use vasopressors, preferably as continuous infusion, for prophylaxis rather than delaying their use until hypotension occurs.

Phenylephrine (PE) is the recommended drug for prophylaxis against hypotension during cesarean delivery; however, the use of PE is commonly associated with decreased heart rate and probably cardiac output because PE is a pure alpha adrenoreceptor agonist. Introduction of NE in obstetric practice had shown favorable maternal and neonatal outcomes and was associated with higher heart rate and cardiac output compared to PE. However, there is still some mothers who develop bradycardia and diminished cardiac output with the use of NE. The most desired scenario during hemodynamic management of mothers during cesarean delivery would achieve the least possible incidences of maternal hypotension, bradycardia and reactive hypertension. Therefore, it is warranted to reach a vasopressor regimen with the most stable hemodynamic profile.

In the last year, epinephrine was reported for the first time in obstetric practice with acceptable safety on the mother and the fetus. However, there is still lack of data about the most appropriate dose for infusion during cesarean delivery. This study aims to compare three prophylactic infusion rates for epinephrine during cesarean delivery.

DETAILED DESCRIPTION:
Upon arrival to the operating room, the patient will be in supine position with left uterine displacement using a wedge below the right buttock. Routine monitoring will be applied (electrocardiography, pulse oximetry, and non-invasive blood pressure monitor). An 18G-cannula will be inserted, and the patients will receive 10 mg metoclopramide. Baseline heart rate and systolic blood pressure will be recorded as the average of three consecutive readings with 2-minutes interval.

Lactated Ringer's solution will be infused at rate of 15 mL/Kg over 10 minutes as a co-load; spinal anesthesia will be achieved by injecting 10 mg of hyperbaric bupivacaine and 20 mcg fentanyl into the subarachnoid space at L3-L4 or L4-L5 interspace using 25G spinal needle.

After subarachnoid block, mothers will be placed in supine position with left-lateral tilt and the vasopressor infusion will be started.

* 0.01 mcg group
* 0.02 mcg group
* 0.03 mcg group The vasopressor infusion will be through the same line as the fluid a three-way stopcock. The vasopressor infusion will be stopped if heart rate became ≥130% of baseline or systolic blood pressure ≥120% of baseline, otherwise the infusion will be stopped 5 minutes after delivery of the baby.

Block success will be assessed after 5 minutes from intrathecal injection of local anesthetic; and will be confirmed if sensory block level is at T4.

Post-spinal hypotension (defined as systolic blood pressure ≤80% of the baseline reading during the period from intrathecal injection to delivery of the fetus) will be managed by administration of 9 mg of ephedrine Severe post-spinal hypotension (defined as systolic blood pressure ≤60% of the baseline reading during the period from intrathecal injection to delivery of the fetus) will be managed by administration IV ephedrine 15 mg.

Reactive hypertension (defined as systolic blood pressure ≥120% of the baseline reading) will be managed by stoppage of the infusion till the next systolic blood pressure reading. The infusion will be then re-started at the half of the initial rate, when systolic blood pressure decreases to be within 20% of the baseline reading.

Intraoperative bradycardia (defined as heart rate less than 55 bpm) will be managed by IV atropine bolus (0.5 mg) will be administered.

Fluid administration will be continued up to a maximum of 1.5 liters. An oxytocin bolus (0.5 IU) will be delivered over five seconds after delivery the infused at a rate of 2.5 IU/hour.

ELIGIBILITY:
Inclusion Criteria:

* full-term singleton pregnant women
* American society of anesthesiologist-physical status I or II,
* scheduled for elective cesarean delivery

Exclusion Criteria:

* Patients with uncontrolled cardiac morbidities (patients with tight valvular lesion, impaired contractility with ejection fraction < 50%, heart block, and arrhythmias),
* hypertensive disorders of pregnancy,
* peripartum bleeding,
* coagulation disorders (patients with INR >1.4 and or platelet count < 80000 /dL) or
* any contraindication to regional anesthesia,
* and baseline systolic blood pressure (SBP) < 100 mmHg

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 276 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
incidence of postspinal hypotension | 1 minute after subarachnoid injection till 5 minutes after baby delivery
  systolic blood pressure ≤80% of the baseline reading

SECONDARY OUTCOMES:
incidence of tachycardia | 1 minute after subarachnoid injection till 5 minutes after baby delivery
  heart rate > 130% of baseline
incidence of hypertension | 1 minute after subarachnoid injection till 5 minutes after baby delivery
  systolic blood pressure >120% of baseline
incidence of severe hypotension | 1 minute after subarachnoid injection till 5 minutes after baby delivery
  systolic blood pressure ≤60% of the baseline reading
mean heart rate | 1 minute after subarachnoid injection, every 2 minutes during procedure, till 5 minutes after baby delivery
  beat per minute
mean systolic blood pressure | 1 minute after subarachnoid injection, every 2 minutes during procedure, till 5 minutes after baby delivery
  mmHg
total ephedrine requirement | 1 minute after subarachnoid injection till 5 minutes after baby delivery
  mg
total atropine requirement | 1 minute after subarachnoid injection till 5 minutes after baby delivery
  mg
Apgar score | 5 minutes after delivery
  Breathing effort Heart rate Muscle tone Reflexes Skin color Each category is scored with 0, 1, or 2, depending on the observed condition
umbilical blood pH | 5 minutes after delivery
  pH
umbilical blood PCO2 | 5 minutes after delivery
  mmHg
umbilical blood PO2 | 5 minutes after delivery
  mmHg
umbilical blood HCO3 | 5 minutes after delivery
  mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Available from PI upon reasonable request

REFERENCES:
- [Derived] Hasanin AM, Abou Amer A, Hassabelnaby YS, Mostafa M, Abdelnasser A, Amin SM, Elsherbiny M, Refaat S. The use of epinephrine infusion for the prevention of spinal hypotension during Caesarean delivery: A randomized controlled dose-finding trial. Anaesth Crit Care Pain Med. 2023 Jun;42(3):101204. doi: 10.1016/j.accpm.2023.101204. Epub 2023 Feb 28. PMID 36858257